CLINICAL TRIAL: NCT07294482
Title: The Effects on Sleep Quality of 1:4 Reishi Liquid Extract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 42486
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single Arm observational where participants act as their own control
  Interventions: Dietary Supplement: Bristol Fungarium's 1:4 Reishi Mushroom Tincture

INTERVENTIONS:
Dietary Supplement: Bristol Fungarium's 1:4 Reishi Mushroom Tincture — UK-grown organic Reishi tincture, cloned in lab. Triple Extracted, 1: 4 Ratio via two hot water extractions and a final organic ethanol extraction to gain access to all the bioactive compounds responsible for Reishi's beneficial properties. (1g of mushrooms to every 4ml of water).

SUMMARY:
Examining the effects of 1ml of Reishi mushroom extract (1:4 extraction ratio, two hot water extractions and an alcohol extraction), taken daily, 30 mins before bed on perceived sleep quality and stress levels. Sleep quality includes: duration, sleep onset latency, nighttime wakings, and perceived restfulness. And consequently, the potential for increased daytime energy levels and a reduction in perceived stress levels.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to meticulously investigate the mythical sleep-enhancing properties of Reishi mushroom, a topic that has garnered significant attention both on social media platforms and in preliminary scholarly research. With a burgeoning interest in natural remedies for sleep disorders and stress management, this study seeks to provide a scientific basis for the anecdotal evidence suggesting the efficacy of Reishi mushroom in these areas. Utilizing a 1:4 Reishi liquid extract, this trial aims to rigorously assess the impact of this ancient remedy on various sleep quality metrics and stress levels among participants.

The core objective of this online study is to offer participants the opportunity to discover personalized insights into how the Reishi tincture influences their sleep patterns and stress levels. By engaging in this research, participants will contribute to a deeper understanding of whether this natural extract can significantly enhance sleep duration, minimize nocturnal awakenings, and elevate overall restfulness, while concurrently reducing stress. This endeavor is geared towards empowering individuals with data-driven results, enabling them to make well-informed decisions regarding their sleep health and lifestyle choices.

In aiming to scientifically evaluate the effects of Reishi extract on sleep quality and stress, participants will receive detailed feedback on how the tincture impacts their unique physiological responses. This personalized approach is intended to assist participants in determining the viability of incorporating such natural supplements into their daily wellness routines.

The significance of this study lies in its potential to challenge and expand current perceptions of natural sleep aids. By substantiating the sleep-enhancing and stress-reducing capabilities of Reishi mushroom, this research could play a pivotal role in revolutionizing how individuals approach their sleep and stress management practices. Although results may vary among participants and certain limitations are to be acknowledged, the study promises to provide valuable, personalized data. This data could significantly influence participants' strategies for achieving restful sleep and effectively managing stress, ultimately contributing to improved daytime energy and overall well-being in a digitally accessible format.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with Allergies
* Pregnant or Nursing Women
* Individuals on Anticoagulants
* Immunocompromised Individuals
* Individuals with Liver Disease
* Children and Adolescents
* Individuals with Chronic Illnesses
* Those with Mental Health Disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (Past Week Version) | Change from baseline (Day 1-5) in perceived stress levels at 4-5 weeks after the start of the intervention
  The Perceived Stress Scale (Past Week Version) is a modified version of the classic stress assessment tool that evaluates stress levels based on recent experiences within the last week. This scale helps in understanding how various situations have recently affected an individual's feelings and perceived stress levels. By focusing on a shorter time frame, it provides a more immediate assessment of stress, which can be particularly useful for quickly evaluating the effectiveness of stress management strategies or interventions. The tool retains its original structure, ensuring its reliability while making it more relevant for current stress evaluation.
  Score Range
  Minimum score: 0
  Maximum score: 40
  Score Interpretation
  Higher scores = worse outcome
  Higher scores indicate greater perceived stress
Neuro-QOL Item Bank v1.0 -Fatigue - Short Form | Change from baseline (Day 1-5) in fatigue levels at 6-7 weeks after the start of the intervention
  This survey aims to assess the level of fatigue experienced by the participant in the past 7 days. Each question should be answered by selecting one of the five options ranging from 'Never' to 'Always'.
  Unabbreviated Scale Title Quality of Life in Neurological Disorders (Neuro-QoL™) Item Bank v1.0 - Fatigue - Short Form
  Score Range
  Raw score range:
  Most commonly used short forms: 8-40
  T-score range (standardized):
  Typically ~30 to ~80, mean = 50, SD = 10
  Score Interpretation
  Higher scores = worse outcome
  Higher scores reflect greater fatigue severity and impact
PROMIS Sleep Disturbance Scale | Change from baseline (Day 1-5) in sleep disturbance levels at 6-7 weeks after the start of the intervention
  The PROMIS Sleep Disturbance Scale is a validated and widely used assessment tool developed as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) initiative. It is designed to measure the severity of sleep disturbances and disruptions experienced by individuals. This scale includes a range of questions that assess the frequency and impact of various sleep-related issues, such as difficulty falling asleep, nighttime awakenings, and restless sleep. Healthcare professionals and researchers rely on this scale to better understand and quantify sleep problems in patients, enabling them to tailor interventions and treatment strategies to address sleep-related concerns effectively.
  Unabbreviated Scale Title Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep Disturbance Scale
  Score Range
  Raw score range:
  6-item short form: 6-30
  Score Interpretation
  Higher scores = worse outcome
  Higher scores indicate greater sleep disturbance (poorer sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=42481